CLINICAL TRIAL: NCT03152617
Title: BASUN - Risks for Malnutrition, Metabolic Bone Disease and Impaired Oral Health After Obesity Treatment - Interaction With Gastrointestinal Microbiota, Psychiatric Morbidity and Socioeconomics
Brief Title: BASUN - Risks for Malnutrition, Metabolic Bone Disease and Impaired Oral Health After Obesity Treatment
Acronym: BASUN
Status: Recruiting | Type: Observational
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: KMossberg
Record Dates: First submitted 2016-10-03; First posted 2017-05-15 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Obesity, Morbid
Keywords: bariatric surgery; gastric bypass; malnutrition; bone disease; oral health
MeSH Terms: conditions — Obesity, Morbid; Malnutrition; Bone Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Weight-reducing obesity surgery (OS) generally gives good results but complications are common; e.g. impaired weight loss, weight regain, bowel pain, diarrhea, vitamin/mineral deficiency, osteoporosis and impaired dental health. The BASUN study is a prospective 10-year comparison of 1000 surgically and 400 conventionally treated individuals regarding adverse side-effects, risk factors for complications and poor outcome.

DETAILED DESCRIPTION:
The use of obesity surgery (OS) has increased dramatically due to the lack of effective conventional weight reducing methods. OS generally gives a sustained weight reduction and improves metabolic co-morbidities but complications are not uncommon, e.g. weight regain, bowel pain, diarrhea, vitamin/mineral deficiency, osteoporosis and impaired dental health. Studies of OS regarding adverse side-effects, risk factors for complications and poor outcomes are few or missing.

The BASUN study is a prospective 10-year comparison of 1000 surgically and 400 conventionally treated individuals. Inclusion started in April 2015 and will be completed in 2017. Subjects are consecutively included from the whole western region of Sweden and are followed by detailed checkups at 2, 5 and 10 years. Protocol includes nutritional and bone status, oral health, psychiatric health, GI symptoms, socioeconomics and health economy. Data are collected by interviews, blood and fecal samples, questionnaires, dual energy x-ray absorptiometry, dentist examinations, patients' record and registries. The study is carried out in close cooperation with experts in surgery, medicine, psychiatry, endocrinology, gastroenterology, hematology, molecular biology, osteoporosis, oral medicine, physiology and general medicine.

The BASUN study will be able to form the basis for more individualized medical guidelines with the objective of improving therapeutic quality and the utilization of health care resources.

ELIGIBILITY:
Inclusion Criteria:

* All patients eligible for obesity treatment under specialist care with medical methods or with surgery

Exclusion Criteria:

* no ability to speak, read or write in Swedish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients eligible for obesity treatment under specialist care with medical methods or with surgery are asked for participation.
Sampling Method: Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2015-04; Primary Completion 2027-04 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Ionized Calcium in serum | 10 years
  Difference between pre- and posttreatment level; unit: mM

SECONDARY OUTCOMES:
Bone mineral density (BMD) | 10 years
  DXA based assessment; units: areal density (g/cm2)
Bone mineral density (T-score) | 10 years
  T-score is bone mineral density (BMD)in relation to young healthy adults of the same sex; unit: number of standard deviations below or above BMD of controls
Bone mineral density (Z-score) | 10 years
  Z-score is bone mineral density (BMD) in relation adults of the same age; unit: number of standard deviations below or above BMD of controls of the same age
Arterial blood pressure | 2, 5 & 10 years
  arterial systolic and diastolic pressure at rest; mmHg
Quality of Life | 2, 5 & 10 years
  36-item Short Form Survey(RAND36); Reported value: reported value: number of (or percentage) patients reporting physical and mental health summary scores indicating moderately to severely reduced quality of life as compared to a general reference population.
Plasma Glucose Concentration | 2, 5 & 10 years
  Fasting value; unit: mM
Serum Insulin Concentration | 2, 5 & 10 years
  Fasting value; unit: mIE/L
Glycated Hemoglobin (HbA1c) | 2, 5 & 10 years
  Unit: mmol/mol
Change in Body Weight From Baseline | 2, 5 & 10 years
  kg
Change in Body Mass Index (BMI) | 2, 5 & 10 years
  kg x m2

OTHER OUTCOMES:
Nutritional status | 2, 5 & 10 years
  Blood biochemistry package: Retinol, RBP, Vitamins B, Vid D, methylmalonate, homocysteine, hemoglobulin, MCV, MCH, MCHC, reticulocytes, iron, transferrin, ferritin , Zn, S-Albumin, creatinine, blood lipid profile, ALP; reported value will be number of patients with one or more abnormal laboratory value(-s).
Psychomorbidity1: Depression | 2, 5 & 10 years
  Patient Health Questionnaire 9 (PHQ-9); reported value: number of (or percentage) patients reporting scores indicating a moderate to severe depressive state
Psychomorbidity2: Anxiety | 2, 5 & 10 years
  Beck Anxiety Inventory (BAI); reported value: number of (or percentage) patients reporting high scores indicating moderate to severe anxiety
Psychomorbidity3: Adult ADHD | 2, 5 & 10 years
  Adult ADHD Self-Report Scale -Screener (ASRS); reported value: number (or percentage) of patients reporting scores above cut-off indicating adult ADHD symptoms
Psychomorbidity4: Drug use | 2, 5 & 10 years
  Drug Use Disorders Identification Test (DUDIT); reported value: number (or percentage) of patients reporting scores above cut-off indicating risk for drug-related problems
Psychomorbidity5: Alcohol | 2, 5 & 10 years
  Alcohol Use Disorders Identification Test (AUDIT); reported value: number (or percentage) of patients reporting scores above cut-off indicating risk for alcohol-related problems
Gastrointestinal symptomatology | 2, 5 & 10 years
  Rome III Diagnostic criteria; reported value: number (or percentage) of patients fulfilling the criteria for functional gastrointestinal gastrointestinal disorder
Oral Health questionnaire | 2, 5 & 10 years
  Oral Health Impact Profile (OHIP-14); reported value: number (or percentage) of patients scoring above cut-off for oral health impacting quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Fandriks, M.D., PhD., Principal Investigator — Institute of Clinical Sciences, the Sahlgrenska Academy, University of Gothenburg
Locations (1):
- Department of Gastrosurgical R & E, the Sahlgrenska Academy,University of Gothenburg, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Celander J, Engstrom M, Hoskuldsdottir G, Lener F, Simons K, Wallenius V, Eliasson B, Hedberg S, Mossberg K. Anaemia and weight outcomes 5 years after metabolic and bariatric surgery - a prospective cohort study. Nutr Metab Cardiovasc Dis. 2025 Dec 11:104521. doi: 10.1016/j.numecd.2025.104521. Online ahead of print. PMID 41486025
- [Derived] Taghat N, Mossberg K, Lingstrom P, Petzold M, Ostberg AL. Impact of Medical and Surgical Obesity Treatment on Dental Caries: A 2-Year Prospective Cohort Study. Caries Res. 2023;57(3):231-242. doi: 10.1159/000533609. Epub 2023 Aug 16. PMID 37586350
- [Derived] Lener F, Hoskuldsdottir G, Landin-Wilhelmsen K, Bjorkelund C, Eliasson B, Fandriks L, Wallenius V, Engstrom M, Mossberg K. Anaemia in patients with self-reported use of iron supplements in the BAriatric surgery SUbstitution and nutrition study: A prospective cohort study. Nutr Metab Cardiovasc Dis. 2023 May;33(5):998-1006. doi: 10.1016/j.numecd.2023.02.008. Epub 2023 Feb 16. PMID 36890072
- [Derived] Taghat N, Lingstrom P, Mossberg K, Fandriks L, Eliasson B, Ostberg AL. Oral health by obesity classification in young obese women - a cross-sectional study. Acta Odontol Scand. 2022 Nov;80(8):596-604. doi: 10.1080/00016357.2022.2063942. Epub 2022 Jul 24. PMID 35876084
- [Derived] Hoskuldsdottir G, Engstrom M, Rawshani A, Lener F, Wallenius V, Fandriks L, Mossberg K, Eliasson B. Comparing effects of obesity treatment with very low energy diet and bariatric surgery after 2 years: a prospective cohort study. BMJ Open. 2022 Apr 8;12(4):e053242. doi: 10.1136/bmjopen-2021-053242. PMID 35396282
- [Derived] Hoskuldsdottir G, Engstrom M, Rawshani A, Wallenius V, Lener F, Fandriks L, Mossberg K, Eliasson B. The BAriatic surgery SUbstitution and nutrition (BASUN) population: a data-driven exploration of predictors for obesity. BMC Endocr Disord. 2021 Sep 10;21(1):183. doi: 10.1186/s12902-021-00849-9. PMID 34507573
- [Derived] Hoskuldsdottir G, Mossberg K, Wallenius V, Al Nimer A, Bjorkvall W, Lundberg S, Behre CJ, Werling M, Eliasson B, Fandriks L. Design and baseline data in the BAriatic surgery SUbstitution and Nutrition study (BASUN): a 10-year prospective cohort study. BMC Endocr Disord. 2020 Feb 14;20(1):23. doi: 10.1186/s12902-020-0503-z. PMID 32059719